CLINICAL TRIAL: NCT04337931
Title: A Phase II Multicenter, Open-label Study to Evaluate the Safety and Efficacy of the CD40 Agonistic Antibody Sotigalimab (APX005M) With or Without Stereotactic Body Radiation Therapy in Adults With Unresectable or Metastatic Melanoma
Brief Title: A Study to Evaluate Sotigalimab (APX005M) in Subjects With Unresectable or Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision (not due to safety reason).
Sponsor: Apexigen America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APX005M-010
Record Dates: First submitted 2020-03-30; First posted 2020-04-08 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Unresectable Melanoma; Metastatic Melanoma; Cancer; Cancer of Skin; Melanoma; Melanoma (Skin)
Keywords: CD40; Immunotherapy; APX005M; sotigalimab
MeSH Terms: conditions — Melanoma; Neoplasms; Skin Neoplasms | interventions — sotigalimab

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be alternately assigned to one of the following 2 cohorts (groups) as long as the cohorts are open:
  Cohort 1: APX005M administered IV at 0.3 mg/kg every 3 weeks (21-day cycle) Cohort 2: APX005M administered IV at 0.3 mg/kg every 2 weeks (14-day cycle) Enrolled participants assigned to Cohorts 1 or 2 that do not receive sotigalimab or are not evaluable for tumor response will be replaced in that cohort before assigning new participants to the other cohort.
  Cohort 3: Participants who have failed any number of prior lines of therapy, sotigalimab administered IV at 0.3 mg/kg in combination with radiation therapy every 2 weeks (14 day cycle) up to 16 weeks followed by sotigalimab administered IV at 0.3 mg/kg every 2 weeks (14-day cycle).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Sotigalimab administered IV at 0.3 mg/kg every 3 weeks (21 day) treatment cycles
  Interventions: Drug: sotigalimab
- Cohort 2 (Experimental): Sotigalimab administered IV at 0.3 mg/kg every 2 weeks (14 day) treatment cycles
  Interventions: Drug: sotigalimab
- Cohort 3 (Experimental): Metastatic melanoma participants who have failed any number of prior lines of therapy with minimum 3 measurable lesions.
  Sotigalimab administered IV at 0.3mg/kg in combination with Stereotactic Body Radiation Therapy (SBRT) every 2 weeks (14-day) treatment cycles up to 16 weeks followed by sotigalimab administered IV at 0.3 mg/kg every 2 weeks (14-day) treatment cycles.
  Interventions: Drug: sotigalimab

INTERVENTIONS:
Drug: sotigalimab — Sotigalimab is a CD40 agonistic monoclonal antibody
  Other Names: APX005M

SUMMARY:
This is a multicenter, open label, Phase 2 study, with 3 parallel cohorts. The aim of the study is to evaluate the efficacy of sotigalimab (APX005M) administered at 2 different schedules to adult participants with unresectable or metastatic melanoma. Participants who have not received prior immunotherapy will be alternately assigned to 1 of 2 cohorts with different sotigalimab administration schedules as long as both are open for enrollment. Participants who have failed any number of prior lines of therapy will be assigned to a 3rd cohort of sotigalimab in combination with radiation therapy.

DETAILED DESCRIPTION:
This is a multicenter, open label, Phase 2 study, with 3 parallel cohorts. The aim of the study is to evaluate the efficacy of Sotigalimab administered at 2 different schedules to adult participants with unresectable or metastatic melanoma who have not received prior immunotherapy. Enrolled participants will be alternately assigned to one of the following 2 cohorts (groups) as long as both cohorts are open.

Cohort 1: APX005M administered IV at 0.3 mg/kg every 3 weeks (21-day cycle) Cohort 2: APX005M administered IV at 0.3 mg/kg every 2 weeks (14-day cycle) Sotigalimab in combination with stereotactic body radiation therapy (SBRT) in adults with unresectable or metastatic melanoma who have failed any number of prior lines of therapy will be assigned to Cohort 3: Sotigalimab administered IV at 0.3 mg/kg in combination with radiation therapy every 2 weeks (14 day cycle) up to 16 weeks followed by sotigalimab administered IV at 0.3 mg/kg every 2 weeks (14-day cycle).

Primary Objective

• Evaluate the overall response rate (ORR) by RECIST 1.1 measurements in each of the cohorts.

Secondary Objectives

* Evaluate the safety of sotigalimab alone or in combination with radiation therapy in each cohort
* Evaluate ORR by modified RECIST 1.1 for immune-based therapeutics (iRECIST) in each cohort
* Evaluate median duration of response (DOR) in each cohort

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable or metastatic melanoma
2. Subjects with BRAF activating mutation must have received a BRAF inhibitor and/or MEK inhibitor regimen prior to study entry
3. Signed written informed consent approved by the relevant local ethics committee(s)
4. Male or female ≥18 years old at time of consent
5. Measurable disease by RECIST 1.1

   a. For Cohort 3 only, subjects must have at least 3 measurable target lesions
6. ECOG performance status of 0 or 1
7. Resolution of all disease or prior treatment-related toxicities to Grade ≤1, with the exception of alopecia, Grade 2 neuropathy and laboratory abnormalities (parameters below apply). If subject received major surgery or radiation therapy of >30 Gy, they must have recovered from the toxicity and/or complications from the intervention
8. Adequate organ function within 14 days prior to first dose of investigational therapy(ies):

   1. WBC ≥2 x 109/L in absence of growth factor support
   2. ANC ≥1.0 x 109/L in absence of growth factor support
   3. Platelet count ≥100 x 109/L
   4. Hemoglobin ≥9 g/dL
   5. Serum creatinine ≤1.5 mg/dL
   6. Calculated (using the formula of local laboratory) or creatinine clearance ≥60 mL/min
   7. AST and ALT ≤2.5 x ULN
   8. Total bilirubin ≤1.5 x ULN, or direct bilirubin ≤ULN with total bilirubin levels >1.5 x ULN
   9. INR or PT ≤1.5 x ULN unless receiving anticoag therapy PT or PTT is within therap, range
   10. aPTT ≤1.5 x ULN unless receiving anticoag therapy PT or PTT is within therap range
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within the 7 days prior to first dose of investigational therapy(ies) and a negative urine pregnancy test within the 3 days prior to first dose of investigational therapy(ies), or a negative serum pregnancy test within the 3 days prior to first dose of investigational therapy(ies)
10. Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of study treatment and 5 months after the last dose of investigational therapy(ies). Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment and 7 months after the last dose of investigational therapy(ies)
11. Available archived or fresh tumor tissue sample for biomarker analysis. Cohort 3, only available archived tissue is required.
12. For subjects that consent to collection of tumor biopsies at study entry and before the first scheduled tumor assessment, primary or metastatic tumor that can be safely biopsied. Up to 18 subjects (6 subjects within each cohort) should consent to fresh core biopsies.

Exclusion Criteria:

1. Prior Therapy:

   1. Cohorts 1 and 2 only: Previous exposure to any immunomodulatory agent (such as CTLA-4, PD-1/PD-L1, IDO inhibitors, interferon, CD40 agonist etc.).
   2. Cohort 3 only: Prior therapy with a CD40 agonist. Any number of prior lines of therapy are eligible. A minimum washout period of 21 days from last line of therapy until investigational therapy(ies) administration should be observed.
2. Second malignancy (solid or hematologic) within the past 3 years except locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
3. Active, known, clinically serious infections (≥ Grade 2 according to NCI-CTCAE v4.03) within the 14 days prior to first dose of investigational therapy(ies)
4. Use of systemic corticosteroids or other systemic immunosuppressive drugs within 28 days prior to first dose of investigational therapy(ies) (except inhaled corticosteroids)

   a. The use of physiologic doses of corticosteroids may be approved /w consultation Medical Monitor (or designee)
5. Major surgery within 4 weeks prior to first dose of sotigalimab
6. Concurrent treatment with any anticancer agent and palliative radiation, unless approved by MM (or designee)
7. History of allogeneic bone marrow transplantation
8. Active, known or suspected autoimmune disease
9. Active autoimmune disease that has required systemic treatment in past 2 years (i.e with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
10. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis
11. History of interstitial lung disease
12. History of sensitivity or allergy to mAbs or IgG
13. Congestive heart failure (New York Heart Association Class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction within 6 months prior to the first dose of investigational therapy(ies)
14. History of any thromboembolic event within 3 months prior to first dose of investigational therapy(ies) or active coagulopathy
15. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with untreated brain metastases ≤3mm that are asymptomatic, do not have significant edema, cause shift, and do not require steroids or anti-seizure medications are eligible after discussion with the Medical Monitor. Lesions of any size in posterior fossa are excluded. Subjects with previously treated brain metastases may participate provided they are stable after treatment (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using corticosteroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
16. Known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection
17. Has received a live (attenuated) vaccine within 30 days prior to the first dose of investigational therapy(ies). Seasonal flu vaccines that do not contain live virus and COVID 19 vaccines are permitted (see Section 3.2.3.4)
18. Has participated in another clinical trial of an investigational drug (or a medical device) within 30 days of study enrollment
19. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
20. Any clinically significant psychiatric, social, or medical condition that, in the opinion of the Investigator, could increase subject's risk, interfere with protocol adherence, or affect a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Poland (2):
  - Szpital Kliniczny im. Heliodora Święcickiego UM w Poznaniu, Poznan
  - Centrum Onkologii - Instytutu im. Marii Skłodowskiej - Curie w Warszawie, Warsaw
- Spain (17):
  - Hospital Universitario San Juan De Alicante, Alicante
  - Hospital Universitari Quirón Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Insular De Gran Canaria, Las Palmas de Gran Canaria
  - Clínica Universidad De Navarra Sede Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen De La Arrixaca, Murcia
  - Hospital Universitario De Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Marqués De Valdecilla, Santander
  - Consorcio Hospital General Universitario de Valenc, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Complexo Hospitalario Universitario De Vigo Álvaro Cunqueiro, Vigo
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 45 participants were enrolled in Poland and Spain between June 2019 and August 2022.
Groups:
- Cohort 1: Participants received 0.3mg/kg of sotigalimab administered intravenously (IV) every 21 days (3 week) treatment cycle.
- Cohort 2: Participants received 0.3mg/kg of sotigalimab administered IV every 14 days (2 week) treatment cycle.
- Cohort 3 -Sotigalimab + Radiation Therapy: Participants received 0.3 mg/kg of sotigalimab administered in combination with stereotactic body radiation therapy (SBRT) every 2 weeks (14-day cycle) up to 16 weeks followed by sotigalimab administered IV at 0.3 mg/kg every 2 weeks (14-day cycle).
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 -Sotigalimab + Radiation Therapy
Started | 12 | 14 | 19
Safety Population | 12 | 13 | 19
Efficacy Population | 11 | 13 | 19
Completed | 0 | 0 | 0
Not Completed | 12 | 14 | 19
Not completed — Death | 4 | 1 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Initiation of subsequent anti-cancer treatment | 1 | 0 | 9
Not completed — Study terminated by sponsor | 3 | 6 | 2
Not completed — Initiated first treatment with anti-PD1/L1 therapy | 3 | 5 | 1
Not completed — Colorectal cancer treatment | 1 | 0 | 0
Not completed — Participant decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population was defined as all participants who received any sotigalimab.
Groups:
- Cohort 1: Participants received 0.3mg/kg of sotigalimab administered IV every 21 days (3 week) treatment cycle.
- Cohort 3: Participants received 0.3mg/kg of sotigalimab administered through IV every 14 days (2 week) treatment cycle in combination with stereotactic body radiation therapy (SBRT) every 14-day cycles (up to 16 weeks) followed by sotigalimab every 14 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 12 | 13 | 19 | 44
Age, Continuous [Median (Full Range); unit: years] | 69.00 [36.00 to 80.00] | 59.00 [40.00 to 85.00] | 63.00 [30.00 to 75.00] | 62.50 [30.00 to 85.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10 | 20
  Male | 8 | 7 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 12 | 10 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 13 | 19 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Poland | 1 | 1 | 8 | 10
  Spain | 11 | 12 | 11 | 34
Weight [Median (Full Range); unit: kg] | 77.20 [51.00 to 96.10] | 79.00 [58.00 to 95.10] | 75.00 [53.00 to 104.00] | 78.10 [51.00 to 104.00]
Height [Median (Full Range); unit: cm] | 169.00 [156.00 to 179.00] | 166.00 [153.00 to 176.00] | 168.00 [146.50 to 185.00] | 168.00 [146.50 to 185.00]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status determines the ability of participants to tolerate therapies in serious illness. 0= Asymptomatic (no symptoms), 1= Symptomatic (exhibits symptoms) but completely ambulatory.
  Participants
    0 (asymptomatic) | 7 | 8 | 7 | 22
    1 (symptomatic but ambulatory) | 5 | 5 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Overall Response Rate (ORR)
Description: The percentage of participants having reached a confirmed Complete Response (CR) or Partial Response (PR) by RECIST 1.1, relative to the number of participants belonging to the Efficacy Population. Confidence Intervals (CIs) were calculated using exact (Clopper-Pearson) method.
  CR: Disappearance of all target lesions and nontarget (NT) lesions; PR: >30% decrease in the sum of the longest diameter of target lesions and no progressive disease in NT lesions or new lesions.
Time Frame: 12 months
Population: Participants evaluable for efficacy (tumor response) are defined as those who have measurable disease and at least one evaluable (post baseline) tumor assessment performed during the treatment period or within 30 days after the administration of the last dose of treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 1: Participants received 0.3mg/kg of sotigalimab administered IV every 21 days (3 week) treatment cycles.
- Cohort 2: Participants received 0.3mg/kg of sotigalimab administered IV every 14 days (2 week) treatment cycles.
- Cohort 3: Participants received 0.3mg/kg of sotigalimab administered IV every 14 days (2 week) treatment cycle in combination with stereotactic body radiation therapy (SBRT) every 14-day cycles (up to 16 weeks) followed by sotigalimab every 14 days.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 19
percentage of participants | 9.09 [0.47 to 36.44] | 7.69 [0.39 to 31.63] | 0.00 [0.00 to 14.59]

2. Secondary Outcome: Modified RECIST 1.1 for Immune-based Therapeutics (iRECIST 1.1) Overall Response Rate (iORR)
Description: The percentage of participants having reached an immune confirmed Complete Response (iCR) or Partial Response (iPR) by iRECIST 1.1, relative to the number of participants belonging to the Efficacy Population. CIs were calculated using exact (Clopper-Pearson) method.
  iCR: Disappearance of all target lesions and NT lesions; iPR: >30% decrease in the sum of the longest diameter of target lesions and no progressive disease in NT lesions or new lesions.
Time Frame: 12 months
Population: iORR for iRECIST 1.1 by Cohort (Efficacy Population).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 3: Participants received 0.3mg/kg of sotigalimab administered IV every 14 days (2 week) treatment cycles in combination with stereotactic body radiation therapy (SBRT) every 14-day cycles (up to 16 weeks) followed by sotigalimab every 14 days.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 19
percentage of participants | 9.09 [0.47 to 36.44] | 7.69 [0.39 to 31.63] | 0.00 [0.00 to 14.59]

3. Other Pre Specified Outcome: RECIST 1.1 Progression-free Survival (PFS)
Description: The PFS was defined as the time (in months) from the first administration of APX005M to the event or censoring date. An event was defined as the first documentation of PD (disease progression assessed based on tumor assessment or clinical progression) or death due to any cause, whichever occurs earlier. Median DoR was calculated using Kaplan-Meier analysis. CIs were calculated using exact (Clopper-Pearson) method.
  PD: >20% increase in the sum of the longest diameter of target lesions and an absolute increase of ≥5mm, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 12 months
Population: PFS for RECIST 1.1 by Cohort (Efficacy Population).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 11 | 13 | 19
months | 1.87 [1.35 to 3.71] | 3.48 [1.81 to 9.20] | 1.87 [1.64 to 1.91]

4. Secondary Outcome: RECIST 1.1 Duration of Response (DoR)
Description: The DoR was defined as the time (in months) from the first evidence of confirmed objective response (CR or PR) to the event or censoring date. An event was defined as the first documentation of progression disease (PD; disease progression assessed based on tumor assessment or clinical progression) or death due to any cause, whichever occurs earlier. Median DoR was calculated using Kaplan-Meier analysis. CIs were calculated using exact (Clopper-Pearson) method.
  CR: Disappearance of all target lesions and NT lesions; PR: >30% decrease in the sum of the longest diameter of target lesions and no progressive disease in NT lesions or new lesions; PD: >20% increase in the sum of the longest diameter of target lesions and an absolute increase of ≥5mm, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 12 months
Population: DoR for RECIST 1.1 by Cohort (Efficacy Population). Inclusive of participants who experienced CR or PR only.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 1 | 1 | 0
months | NA [NA to NA] — Median and CIs were not reached due to low number of events | NA [NA to NA] — Median and CIs were not reached due to low number of events |

ADVERSE EVENTS:
Time Frame: Up to approximately 79 weeks
Description: All AE's below are reported regardless of relationship to treatment.
Groups:
- Cohort 1: Sotigalimab infusion (IV) 0.3 mg/kg every 3 weeks (21 day) treatment cycles.
- Cohort 2: Sotigalimab infusion (IV) 0.3 mg/kg every 2 weeks (14 day) treatment cycles.
- Cohort 3: Sotigalimab infusion (IV) 0.3 mg/kg every 2 weeks (14 day) treatment cycle plus Stereotactic Body Radiation Therapy (SBRT) every 14 day-cycles (up to 16 weeks) followed by sotigalimab every 14 days in adults with unresectable or metastatic melanoma who have failed any number of prior lines of therapy.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 4/12 | 1/13 | 7/19
Serious Adverse Events (participants affected / at risk) | 7/12 | 0/13 | 3/19
Other Adverse Events (participants affected / at risk) | 12/12 | 12/13 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=13) | Cohort 3 (N=19)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=12) | Cohort 2 (N=13) | Cohort 3 (N=19)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 4 (7)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (13) | 4 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (10) | 1 (1)
Asthenia (General disorders) | 4 (4) | 7 (11) | 4 (4)
Chills (General disorders) | 2 (2) | 6 (7) | 5 (6)
Pyrexia (General disorders) | 7 (17) | 7 (15) | 13 (20)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (4) | 4 (5) | 2 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 8 (11)
Alanine aminotransferase increased (Investigations) | 6 (13) | 6 (14) | 7 (9)
Aspartate aminotransferase increased (Investigations) | 7 (12) | 6 (10) | 8 (11)
Blood creatinine increased (Investigations) | 2 (3) | 3 (4) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 4 (6) | 3 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (7) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 3 (3)
Hypertension (Vascular disorders) | 1 (1) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 4 (5)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 2 (4) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 2 (4) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Uticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04337931/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04337931/SAP_001.pdf